CLINICAL TRIAL: NCT03018574
Title: Candidate Gene Screening for 6-14 Year Old Patients With ADHD (Attention Deficit/ Hyperactivity Disorder)
Brief Title: Candidate Gene Screening for Attention Deficit/Hyperactive Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20163381
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2017-01

CONDITIONS: Gene Product Sequence Variation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD-patients: The whole blood sample from diagnoses of the children 6-14 years old with ADHD. Diagnoses of the children with ADHD were made in Xijing Hospital and Children's Hospital Affiliated to Soochow University according to criteria described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Children with ADHD had an IQ score above 70.
- Controls-healthy children: The whole blood sample from age- and gender- matched healthy 6-14 years old children

SUMMARY:
Source: Sample bank of Xijing Hospital and Children's Hospital Affiliated to Soochow University; Sample form: Whole blood; Estimated number of samples: 100 patients with ADHD and age, sex matched healthy controls; Case exclusion criteria: all kinds of neuropsychiatric disorders, IQ value of less than 70;

Study protocol:

1. Using Qiagen kit to extract the genomic DNA of 200 microliters of blood.
2. UV spectrophotometer test DNA purity of 260/280 close to 1.8 (1.8 ± 0.05), the concentration of 100ng/μL or more before the next sequencing.
3. The extracted genomic DNA will be sent to Sangon Biology Engineering Limited Company (Shanghai) and sequenced to find candidate mutations related to ADHD risk sequence. According to NIH gene database, the longest transcript of NDRG2 (ID: 57447 gene, https://www.ncbi.nlm.nih.gov/nuccore/NC_000014.9? Report=genbank&from=21016763&to=21070872&strand=true) (a total of 17 exons and 16 introns and the gene 5 'UTR and 3' UTR region) will be alignmented sequences to find potential mutations.
4. Using the chi square analysis and other statistical methods to determine the relationship between the mutations and susceptibility to ADHD.

DETAILED DESCRIPTION:
Source: Sample bank of Xijing Hospital and Children's Hospital Affiliated to Soochow University; Sample form: Whole blood; Estimated number of samples: 100 patients with ADHD and age, sex matched healthy controls; Case exclusion criteria: all kinds of neuropsychiatric disorders, IQ value of less than 70;

Study protocol:

1. Using Qiagen kit to extract the genomic DNA of 200 microliters of blood. (1) melt frozen blood at room temperature; (2) take the blood of 0.2 ml into a sterile anti coagulation centrifuge tube, add an equal volume of PBS phosphate buffer, after fully mixing 12000rpm centrifugation 5min, discard supernatant; (3) 66.7 L STE 2.4 L, 20% SDS, 37 DEG C water bath 1h; (4) protease K plus 1 20mg/ml l mix, 55 DEG C water bath digestion overnight (10 ~ 14h); (5) the digested samples treated with Tris saturated phenol, shake well, 12000rpm centrifugal 10min; (6) the upper aqueous phase to a sterile centrifuge tube; adding volume of Tris saturated phenol, shake well, 12000rpm centrifugal 10min; (7) the upper aqueous phase was transferred to another sterile centrifuge tube, and an equal volume of phenol was added: chloroform: isoamyl alcohol (25: 24: 1). The oscillation of the vortex was fully mixed, and the 12000rpm was centrifuged to 10min; (8) the upper aqueous phase was transferred to another sterile centrifuge tube, and an equal volume of chloroform was added: iso amyl alcohol (24: 1), which was fully vibrated and mixed with 12000rpm centrifugation 10min; (9) transfer the supernatant to another sterile centrifuge tube; adding 2 times volume ethanol, the volume level of sodium acetate 1/10 shake, until the flocculent precipitation of DNA visible; (10) the sample is placed at -20 DEG C refrigerator freezer 30min or ice bath for 15 ~ 20min, after removal of 12000rpm centrifugal 10min again, so that DNA precipitation; (11) the gun head will pick DNA to another sterile centrifugal tube, with the amount of 70% ethanol washing and shaking, to wash out impurities DNA; (12) out of ethanol, DNA by vacuum drying or dry naturally, TE buffer adding dissolution, -20 stored at standby.
2. UV spectrophotometer test DNA purity of 260/280 close to 1.8 (1.8 ± 0.05), the concentration of 100ng/μL or more before the next sequencing.
3. The extracted genomic DNA will be sent to Sangon Biology Engineering Limited Company (Shanghai) and sequenced to find candidate mutations related to ADHD risk sequence. According to NIH gene database, the longest transcript of NDRG2 (ID: 57447 gene, https://www.ncbi.nlm.nih.gov/nuccore/NC_000014.9? Report=genbank&from=21016763&to=21070872&strand=true) (a total of 17 exons and 16 introns and the gene 5 'UTR and 3' UTR region) will be alignmented sequences to find potential mutations.
4. Using the chi square analysis and other statistical methods to determine the relationship between the mutations and susceptibility to ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of the children with ADHD were made in Xijing Hospital and Children's Hospital Affiliated to Soochow University according to criteria described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Children with ADHD had an IQ score above 70.

Exclusion Criteria:

* Children who had a past history of or were currently affected by neurological diseases, including convulsive disorders or brain damage; or who had any evidence of comorbid psychiatric conditions, such as Tourette's syndrome, IQ below 70, pervasive developmental disorder (autism), bipolar disorder, psychosis, language difficulties or learning disorders (reading disorders, mathematics disorders and disorders of written expression).

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Diagnoses of the children with ADHD were made in Xijing Hospital and Children's Hospital Affiliated to Soochow University according to criteria described in the Diagnostic and Statistical Manual of Mental Disorders. Children with ADHD had an IQ score above 70.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Gene point mutation in the genome of ADHD patients and healthy controls | 2016-2017

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, PhD&MD, Principal Investigator — Xijing hospital of The fourth military medical university
Locations (1):
- Xijing Hospital of the Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Publish all data in a paper

REFERENCES:
- [Result] Won H, Mah W, Kim E, Kim JW, Hahm EK, Kim MH, Cho S, Kim J, Jang H, Cho SC, Kim BN, Shin MS, Seo J, Jeong J, Choi SY, Kim D, Kang C, Kim E. GIT1 is associated with ADHD in humans and ADHD-like behaviors in mice. Nat Med. 2011 May;17(5):566-72. doi: 10.1038/nm.2330. Epub 2011 Apr 17. PMID 21499268
- [Result] Salatino-Oliveira A, Genro JP, Chazan R, Zeni C, Schmitz M, Polanczyk G, Roman T, Rohde LA, Hutz MH. Association study of GIT1 gene with attention-deficit hyperactivity disorder in Brazilian children and adolescents. Genes Brain Behav. 2012 Oct;11(7):864-8. doi: 10.1111/j.1601-183X.2012.00835.x. Epub 2012 Sep 7. PMID 22897819
- [Result] Vegt R, Bertoli-Avella AM, Tulen JH, de Graaf B, Verkerk AJ, Vervoort J, Twigt CM, Maat-Kievit A, van Tuijl R, van der Lijn M, Hengeveld MW, Oostra BA. Genome-wide linkage analysis in a Dutch multigenerational family with attention deficit hyperactivity disorder. Eur J Hum Genet. 2010 Feb;18(2):206-11. doi: 10.1038/ejhg.2009.148. Epub 2009 Aug 26. PMID 19707245